CLINICAL TRIAL: NCT03796832
Title: The FiREwORK Trial - Self-management With FootweaR Combined With Exercise for OsteoaRthritis (OA) at the Knee: a Phase II Randomized Controlled Trial
Brief Title: Footwear and Exercise for Knee Osteoarthritis (FiREwORK Trial)
Acronym: FiREwORK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B670201835057; G013318N (Other Grant/Funding Number: Fonds voor Wetenschappelijk Onderzoek (FWO)); U1111-1225-9954 (Other: WHO)
Record Dates: First submitted 2018-12-21; First posted 2019-01-08 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Exercise Therapy; Shoes; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: This will be a mono-centre randomized controlled trial with a 1:1 allocation into the experimental treatment (exercise therapy and Flat Flexible Shoes) and comparator treatment (exercise therapy and Stable Supportive Shoes). Exercise therapy will consist of supervised facility- and home-based exercises for 3 months (primary time point) and unsupervised home-based exercises for a subsequent 6 months (secondary time point).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flat Flexible Shoes+Exercise Therapy (Experimental): This arm will wear Flat Flexible Shoes daily for the duration of 9 months combined with supervised facility-based and home-based exercise therapy (months 0-3) and unsupervised home-based exercise therapy (months 4-9).
  Interventions: Device: Flat Flexible Shoes; Other: Exercise Therapy
- Stable Supportive Shoes+Exercise Therapy (Active Comparator): This arm will wear Stable Supportive Shoes daily for the duration of 9 months combined with supervised facility-based and home-based exercise therapy (months 0-3) and unsupervised home-based exercise therapy (months 4-9).
  Interventions: Device: Stable Supportive Shoes; Other: Exercise Therapy

INTERVENTIONS:
Device: Flat Flexible Shoes — Off-the-shelf commercially available shoes will be used compliant with previously published criteria: (i) heel height <15 mm, (ii) shoe pitch <10 mm, (iii) absent arch support/motion control, (iv) minimal sole rigidity, (v) weight <=200g (+/-10%). Participants will be instructed to wear the shoes at least 4 hours daily for the duration of the 9-month intervention and to avoid wearing other types of shoes, if possible.
  Arms: Flat Flexible Shoes+Exercise Therapy
Device: Stable Supportive Shoes — Off-the-shelf commercially available shoes will be used compliant with previously published criteria: (i) heel height >30 mm, (ii) shoe pitch >10 mm, (iii) present arch support/motion control, (iv) sole rigidity, (v) weight >300g (+/-10%). Participants will be instructed to wear the shoes at least 4 hours daily for the duration of the 9-month intervention and to avoid wearing other types of shoes, if possible.
  Arms: Stable Supportive Shoes+Exercise Therapy
Other: Exercise Therapy — The 3-month supervised exercise program will consist of one group session per week of approximately 30 minutes complemented with home-based exercises 3 times per week. Group sessions will consist of a 10-min warm-up followed by a circuit training of strengthening and/or neuromuscular exercises. Subsequently, during a 6-month unsupervised home exercise program, participants will perform strengthening exercises of the lower limb muscles 3 times weekly. Throughout the 9-month intervention, participants will be encouraged to maintain a daily routine of aerobic exercises, consisting of structured activity bouts of at least 10 minutes at a moderate intensity (grade 5-6 (out of 10, maximum exertion) on a Rate of Perceived Exertion scale), achieving at least 70 minutes of weekly physical activity at 3 months and 150 minutes at 9 months.

SUMMARY:
Osteoarthritis (OA) is a chronic degenerative joint disease and leading cause of musculoskeletal pain and disability worldwide. The high rates of knee replacement surgery worldwide emphasize the need for more effective non-surgical interventions to attenuate progressive disability. International scientific and professional societies also propose that therapies need to seek efficacious combinations of modalities with the ultimate aim to achieve longer-term, optimal and synergistic treatment effects.

Exercise therapy, such as strengthening and aerobic exercise, is universally, and strongly, recommended as it demonstrates beneficial effects on clinical symptoms and is considered safe for all patients with knee OA. However, during activities as simple as walking, higher knee joint loads have been demonstrated in people with medial tibiofemoral OA, a common form of knee OA. Increased joint loading as such may elicit aggravated symptoms and accelerated joint structural decline over time. No convincing evidence exists to confirm exercise therapy effectively alters joint loading parameters during walking gait in people with knee OA. Notably, recent studies suggest that wearing appropriate footwear may help offload the joint in people with knee OA, a strategy that is also easily applicable at a wide population level.

The purpose of this clinical study is to compare 9-month treatment consisting of exercise therapy and daily wear of one of two shoe classes (flat flexible shoes or stable supportive shoes), on symptom relief and joint structural damage in people with knee OA. In this study, we will randomly allocate eligible participants in one of two treatment arms. This means there will be an equal amount of participants in each group, and participants nor researchers will be able to choose in which group participants will end up in.Participants in both groups will enroll in a 9 month exercise program and will be provided a pair of one of the two shoe classes to wear daily. To ensure an unbiased appraisal of treatment effects, we will not disclose the study hypotheses to participants during the intervention period.

The results of this study will help determine whether the addition of appropriate footwear to exercise therapy improves symptom relief and/or slows structural disease progression in people with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic and radiographic diagnosis of knee OA as per the American College of Rheumatology criteria (ie, aged≥50, knee pain on most days and osteophytes)
* Radiographic evidence of medial OA (ie, Kellgren Lawrence(KL) grade ≥2, ≥grade 1 medial joint space narrowing (JSN) (scale 0-3)> lateral JSN, using a standardized atlas)
* Average knee pain on walking over the past week of ≥4 on a 11-point numeric rating scale (NRS; "0=no pain" to "10=worst pain imaginable")
* Ability to walk unaided
* Willing to comply with therapy prescriptions
* Sufficient understanding of the Dutch language

Exclusion Criteria:

* Current and previous (3 months) participation in exercise therapy
* Current and previous (3 months) use of customised footwear, minimalist shoes, insoles, braces and unable/unwilling to abandon during the study
* Knee surgery in either knee and/or injections (corticosteroids, hyaluronic acid) in the study knee (most painful knee or right knee if both equally painful) in the past 6 months
* Current or recent (4 weeks) use of oral corticosteroids
* Knee replacement or high tibial osteotomy surgery in the past, or planned during the study
* Inflammatory arthropathies
* Other muscular, joint, neurological or metabolic conditions affecting lower limb function and/or precluding safe regular participation in exercise therapy and walking
* Body mass index (BMI) of >36 kg/m2 (due to difficulties performing gait analysis and MRI)
* Foot/ankle pain/pathologies at either side, and worse than knee pain complaints
* Contra-indications for radiography & MRI
* Use of supplements (eg, glucosamine, chondroitin, curcuma derivates) or pain medication (NSAIDs, paracetamol) or other disease modifying or anti-bone resorptive drugs if participants were not on a stable dose for ≥2 months prior to entering the trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change in severity of knee pain on walking | Measured at baseline, 13 and 37 weeks
  Scored on an 11-point numeric rating scale for average knee pain on walking over the past week, with terminal descriptors of "0=no pain" to "10=worst pain imaginable".

SECONDARY OUTCOMES:
Severity of intercondylar synovitis | Measured at baseline, 13 and 37 weeks
  Graded using the MRI Osteoarthritis Knee Score hoffa-synovitis sub-score, ranging grade 0 (normal) to grade 3 (severe).
Severity of whole knee effusion | Measured at baseline, 13 and 37 weeks
  Graded using the MRI Osteoarthritis Knee Score effusion-synovitis sub-score, ranging grade 0 (physiologic amount) to grade 3 (large - evidence of capsular distention).
Severity of bone marrow lesions | Measured at baseline, 13 and 37 weeks
  Graded using the MRI Osteoarthritis Knee Score bone marrow lesion sub-score, grade 0 (none) to grade 3 (>66% of subregional volume).
Severity of physical dysfunction | Measured at baseline, 13 and 37 weeks
  Measured with the function subscale of the Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index. This sub-scale gives a range of possible scores from "0=no dysfunction" to "68=maximum dysfunction".
Severity of knee pain overall | Measured at baseline, 13 and 37 weeks
  Scored on an 11-point numeric rating scale for average knee pain overall the past week, with terminal descriptors of "0=no pain" to "10=worst pain imaginable".
Participant-perceived global change in pain | Measured at 13 and 37 weeks
  Scored on a 7-point ordinal scale (with terminal descriptors of "1=much worse" to "7=much better"). Participants who report they are "moderately better" and above will be classified as "improved".
Participant-perceived global change in physical function | Measured at 13 and 37 weeks
  Scored on a 7-point ordinal scale (with terminal descriptors of "1=much worse" to "7=much better"). Participants who report they are "moderately better" and above will be classified as "improved".
Participant-perceived global change overall | Measured at 13 and 37 weeks
  Scored on a 7-point ordinal scale (with terminal descriptors of "1=much worse" to "7=much better"). Participants who report they are "moderately better" and above will be classified as "improved".
Average Daily Step Count | Measured during weeks 1, 12 and 36
  Measured using a pedometer attached to the hip for 7 subsequent days to assess objective physical activity.
Habitual physical activity level | Measured at baseline, 13 and 37 weeks
  Measured using the Physical Activity Scale for the Elderly with scores ranging 0-400 where higher scores indicate greater physical activity.
Health-related quality of life | Measured at baseline, 13 and 37 weeks
  Measured using the EuroQoL Quality of Life Scale (EQ-5D) with scores ranging from 0 to 100 (higher scores indication better health-related quality of life).

OTHER OUTCOMES:
Adherence to shoe usage | Measured by pedometer at week 1, week 12, week 37, and by logbooks at month 1 , month 2, month 3, month 4, month 5, month 6, month 7, month 8, month 9
  Measured using a shoe-mounted pedometer on week 1, 12 and 37 for 7 consecutive days and by self-report in logbooks for one week during each month. The number of hours of daily shoe wearing will be recorded for 7 consecutive days and compliance will be rated using an 11-point NRS (with terminal descriptors "0=never worn" to "10=always worn").
Adherence to exercise therapy | Measured at week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12 and month 4, month 5, month 6, month 7, month 8, month 9
  During the supervised 12-week phase, participants will record completed exercise sessions every week in a logbook and will complete weekly 11-point NRS scales rating their overall compliance with the exercise prescription (with terminal descriptors: "0= not at all compliant" to "10=extremely compliant"). Therapists will record participants' attendance. During the 6-month phase, patient-reported adherence will be collected for one week each month.
Adverse events, co-interventions including medication use | Measured at baseline, 13 and 37 weeks
  will be collected monthly using logbooks and will also be quired by questionnaire.
Knee joint loading - lower limb kinetics and kinematics | Measured at baseline, 13 and 37 weeks
  An 8-camera optical motion capture system and a force plate will be used to collect kinematic and ground reaction forces. Participants will perform barefoot walking trials at a self-selected walking speed until seven complete "clean" foot strikes (satisfactory force plate contact defined as initial contact at the heel and toe off occurring on the force plate)) will be recorded from both limbs. At 36 weeks, participants will perform gait analysis under two conditions (in random order): (i) barefoot and (ii) allocated shoe. Major parameters of interest will be: (i) peak knee adduction moment, (ii) knee adduction moment angular impulse, and (iii) peak knee flexion moment. Unblinded scientific personnel and a blinded PhD student will collect the gait data. At 36 weeks the PhD student will be unblinded during the 3D gait analyses (last test of the testing session). Subsequent analyses will be performed by the blinded PhD student.
Markers of local synovial inflammation - synovial hypertrophy and Doppler activity | Measured at baseline, 13 and 37 weeks
  Will be measured using an ultrasound machine with a 10-18 MHz linear array transducer. The regions examined will be: the suprapatellar recess, the medial and lateral parapatellar recesses and the medial and lateral femorotibial joint space. All anterior scans will be performed in the longitudinal position except for the parapatellar recess (transverse). Posteriorly, The medial aspect of the popliteal space will be assessed both in the longitudinal and transversal position to assess Baker's cyst presence. All US examinations will be carried out by one unblinded investigator with the participant lying supine on an examination table (knee flexed to 30°), except for the Baker's cyst assessment in which the participant is prone (knee fully extended). The same investigator will evaluate all images for capsular distension, synovial Doppler activity, synovial hypertrophy, effusion and presence of Baker's cyst. The investigator will be blinded to participant ID and test date.
Neuropathic pain | Measured at baseline, 13 and 37 weeks
  Will be assessed using the modified painDETECT questionnaire (mPDQ) a 12-item patient-based, screening questionnaire to determine the presence of neuropathic pain components validated in a range of conditions including OA.
Foot posture | Measured at baseline, 13 and 37 weeks
  Will be assessed using the Foot Posture Index (FPI), a valid and reliable tool that scores six features of foot posture from - 2 (more supinated) to + 2 (more pronated).
Location of knee pain | Measured at baseline, 13 and 37 weeks
  The Photographic Knee Pain Map will be used to determine location of knee pain. The map consists of a photographic representation of the anterior view of a pair of knees on which the participant can mark all painful locations in their study knee.
Numbers of participants dropped out from study | From baseline to 9 months
  Participants who will stop participating in the study (either due to loss to follow-up or study withdrawal) will be asked by mail or telephone to provide the reason why they dropped out from the study. These information will be formally recorded throughout the trial by the trial coordinator.
Peripheral sensitization (thermal) | Measured at baseline, 13 and 37 weeks
  Will be measured assessing heat detection and pain thresholds on the study knee (i.e., most painful knee) by one (always the same) blinded investigator.Heat contact thermal stimuli will be delivered using a computer-controlled (Medoc Pathway Pain & Sensory Evaluation System).
Widespread sensitization (thermal) | Measured at baseline, 13 and 37 weeks
  Will be measured assessing heat detection and pain threshold on a remote peripheral site (i.e., extensor carpi radialis longus) by one (always the same) blinded investigator. Heat contact thermal stimuli will be delivered using a computer-controlled (Medoc Pathway Pain & Sensory Evaluation System).
Pain sensitivity (local) | Measured at baseline, 13 and 37 weeks
  Will be measured by temporal summation (TS) at the study knee (i.e., most painful knee) performed by one (always the same) blinded investigator. Heat contact thermal stimuli will be delivered using a computer-controlled (Medoc Pathway Pain & Sensory Evaluation System). Heat stimuli will be individualized for each subject. Participants will receive10 heat pulses. Participants will be asked to provide a verbal pain rating on a 11-point (0-10) numeric rating scale (NRS) (0 = no pain and 10 = most intense pain imaginable) at 1st; 5th and 10th pulse. TS will be derived according to established protocols.
Pain sensitivity (peripheral) | Measured at baseline, 13 and 37 weeks
  Will be measured by temporal summation (TS) on a remote peripheral site (i.e., extensor carpi radialis longus) performed by one (always the same person) blinded investigator. Heat contact thermal stimuli will be delivered using a computer-controlled (Medoc Pathway Pain & Sensory Evaluation System). Heat stimuli will be individualized for each subject. Participants will receive10 heat pulses. Participants will be asked to provide a verbal pain rating on a 11-point (0-10) numeric rating scale (NRS) (0 = no pain and 10 = most intense pain imaginable) at 1st; 5th and 10th pulse. TS will be derived according to established protocols.
Peripheral sensitization (mechanical) | Measured at baseline, 13 and 37 weeks
  Pressure pain thresholds (PPTs) will be performed on the study knee (i.e., most painful knee) by eliciting mechanical pressure pain applied perpendicular to the skin using an analogue algometer. PPTs will be performed by one (always the same person) blinded investigator.
Widespread sensitization (mechanical) | Measured at baseline, 13 and 37 weeks
  Pressure pain thresholds (PPTs) will be performed on a remote peripheral site (i.e., extensor carpi radialis longus) by eliciting mechanical pressure pain applied perpendicular to the skin using an analogue algometer. PPTs will be performed by one (always the same person) blinded investigator.
Dysfunctional endogenous analgesia | Measured at baseline, 13 and 37 weeks
  Will be assessed by conditioned pain modulation (CPM) at the study knee (i.e., most painful knee) by one (always the same person) blinded investigator. CPM will be measured using a test stimulus followed by a conditioning stimulus and re-assessment of the test stimulus during and after the conditioning stimulus.
Dysfunctional endogenous analgesia | Measured at baseline, 13 and 37 weeks
  Will be assessed by conditioned pain modulation (CPM) on a remote peripheral site (i.e., extensor carpi radialis longus) by one (always the same person) blinded investigator. CPM will be measured using a test stimulus followed by a conditioning stimulus and re-assessment of the test stimulus during and after the conditioning stimulus.
Central sensitization | Measured at baseline, 13 and 37 weeks
  Will be assessed using the central sensitisation inventory (CSI).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Calders, PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Department of Rehabilitation Sciences, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dainese P, Stautemas J, De Mits S, Wittoek R, Van Ginckel A, Huysse W, Demeyer H, Mahieu H, Calders P. Exercise and footwear in medial knee osteoarthritis: a randomized controlled trial comparing flat flexible footwear to stable supportive shoes. Rheumatol Adv Pract. 2024 Oct 30;8(4):rkae133. doi: 10.1093/rap/rkae133. eCollection 2024. PMID 39669115